CLINICAL TRIAL: NCT00572936
Title: Circadian Rhythms of Aqueous Humor Dynamics in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0405-05-FB
Record Dates: First submitted 2007-12-07; First posted 2007-12-13 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Glaucoma
Keywords: Glaucoma; Ocular Hypertension; Timolol®, Latanoprost® and Dorzolamide®
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost; dorzolamide; Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Latanoprost/Dorzolamide/Timolol (Other): The participants received latanoprost at night and vehicle in the morning for two weeks, then 6 week washout, then Dorzolamide BID for two weeks, then 6 week washout, then Timolol BID for two weeks. The order in which the participants received the three different drugs was random.
  Interventions: Drug: Latanoprost; Drug: Dorzolamide; Drug: Timolol

INTERVENTIONS:
Drug: Latanoprost — prostaglandin
  Other Names: xalatan
Drug: Dorzolamide — carbonic anhydrase inhibitor
  Other Names: trusopt
Drug: Timolol — beta blocker
  Other Names: Timoptic, Betimol, Timoptic-xe, Istalol, Timoptic Ocudose

SUMMARY:
This study is designed to identify physiological, pharmacological and pathological circadian fluctuations in aqueous humor inflow and outflow, systemic blood pressure and ocular blood flow in humans.

DETAILED DESCRIPTION:
Glaucoma is a progressive optic neuropathy and a leading cause of blindness in the United States. In glaucoma, vision is lost through apoptosis (programmed cell death) of retinal ganglion cells, a type of cell in the retina that transmits visual information to the brain. Diagnosis of glaucoma is usually based on a combination of progressive, characteristic vision loss (measured using visual field testing) and progressive optic nerve head damage (as detected through dilated fundus examinations or disc photography). While a high pressure inside the eye (ocular hypertension, OHT) is not sufficient for a diagnosis of glaucoma, it is the greatest single risk factor for disease onset.

Currently, the only effective treatment to prevent disease progression is lowering of the intraocular pressure (IOP). IOP is determined by the balance between aqueous production (flow) and aqueous outflow through either the trabecular meshwork or uveoscleral pathway. Diurnal rhythms in aqueous humor dynamics and nocturnal fluctuations in IOP and aqueous flow have been studied in some detail9 but little is known about the nocturnal rhythms of aqueous humor outflow.

Usually, clinical IOP measurement is performed during the day; little is known about nocturnal IOP fluctuations in relation to glaucoma management . A recent surge of interest in nocturnal IOPs stems from the hypothesis that significant glaucomatous damage may occur at night. In response, some investigators have advocated particular classes of glaucoma medications based on their nocturnal IOP effects. The most efficacious drug on the market may not be the preferred treatment if it is ineffective at night. Therefore, the understanding of nighttime IOP and the aqueous humor dynamics that control it has important scientific, clinical, and commercial implications.

Additionally, previous research on glaucoma medications has been limited to the effects ocular hypotensive drugs on 24-hour IOP or daytime aqueous humor dynamics; few studies have addressed their effect on nocturnal aqueous humor dynamics. Beta-blockers have been proven effective in lowering IOP during the day by decreasing aqueous flow. However, limitations have been found in their IOP-lowering effect overnight. Prostaglandins, which increase uveoscleral outflow, seem to possess a hypotensive effect that is constant throughout the 24-hour period. Dorzolamide reduces aqueous flow to lower IOP but few studies have addressed its effect at night. This study is designed to elucidate the physiological mechanisms driving the efficacy of these drugs throughout the 24-hour period, i.e. circadian rhythms in aqueous humor dynamics.

In studies of new glaucoma medications the preferred study population includes ocular hypertensive subjects. These people have high IOP but no optic nerve damage and no glaucoma. They may be taking prescribed IOP lowering drugs for this condition or they may not. Those taking ocular drugs are asked to stop taking them. Since each of the glaucoma drugs affects aqueous humor dynamics in different ways, it is essential that no residual medical effect remains from these drugs. Standard washout periods of 6-weeks will be utilized in between drug assessments. This period of time is based on the methods of other published studies which determined a necessary period of 4-8 weeks for ocular washout of prostaglandins. A concern for patient safety exists when OHT patients are taken off of glaucoma medications, as IOP may rise during the washout. In order to monitor IOP in these patients, most study methods utilize a biweekly check of the IOP. If pressure rises above the ophthalmologist's preset "target pressure" at any point, then the patient is removed from the study and returned to their previous medical regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be nineteen (19) years of age or older. Subjects must be able and willing to give written informed consent [i.e., each subject will be given ample time to read (or have read to them) the consent form, ask any questions they may have regarding the study, and have a clear understanding of the study as well as the procedures involved, prior to signing the consent form].
* Subjects must exhibit a willingness to comply with the protocol and investigator's instructions.
* Subjects must have been previously diagnosed with unilateral or bilateral ocular hypertension at least six months prior to the screening visit.
* Subjects must exhibit baseline IOPs between 21 and 35 mmHg (inclusive); the average IOP between eyes must be ≤ 5 mmHg
* Subjects will be age matched to ocular hypotensive subjects
* Subjects must exhibit baseline IOPs between 12 and 20 mmHg (inclusive); the average IOP between eyes must be ≤ 5 mmHg

Exclusion Criteria:

* Age less than nineteen years old.
* Women who are pregnant, lactating or of childbearing potential who are not using highly effective birth control measures.
* Aphakia or pseudophakia
* Best corrected visual acuity worse than 20/60 in either eye.
* Chronic or recurrent severe ocular inflammatory disease.
* Ocular infection or inflammation within three (3) months of screening visit.
* History of clinically significant or progressive retinal disease such as retinal degeneration, diabetic retinopathy or retinal detachment.
* Any abnormality preventing reliable tonometry of either eye.
* Previous exposure to: beta-adrenergic antagonists, topical prostaglandin analogues (including latanoprost, unoprostone, travoprost and bimatoprost) within six (6) weeks of the baseline visit; α-adrenergic agonists within two (2) weeks of the baseline visit; and cholinergic agonists and carbonic anhydrase inhibitors within five (5) days of the treatment initiation visit
* History of any severe ocular pathology (including severe dry eye) that would preclude the administration of a topical beta blocker, carbonic anhydrase inhibitor, or a topical prostaglandin.
* Any eye with a cup-to-disc ratio greater than 0.8.
* History of intraocular surgery.
* History of ocular laser surgery.
* History of severe or serious hypersensitivity to topical or systemic beta blockers, prostaglandins, or sulfa drugs.
* History of severe, unstable or uncontrolled cardiovascular, hepatic or renal disease.
* History of bronchial asthma or chronic obstructive pulmonary disease (COPD).
* Less than one month (prior to baseline) stable dosing regimen of any non-glaucoma medication that would affect IOP.
* Gonioscopy angle < 2.
* Inability to be dosed with treatment medication.
* Inability to discontinue contact lens wear.
* Therapy with any investigational agent within 30 days of screening.
* Use of any additional topical or systemic adjunctive ocular hypotensive medications during the study.
* History of open angle glaucoma (either primary open angle glaucoma or other cause of open angle glaucoma) or narrow angle glaucoma.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-03-13 (Actual); Primary Completion 2009-11-01 (Actual); Study Completion 2009-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl B Camras, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Department of Ophthalmolgy and Visual Sciences, Omaha, Nebraska, United States

REFERENCES:
- [Result] Gulati V, Fan S, Zhao M, Maslonka MA, Gangahar C, Toris CB. Diurnal and nocturnal variations in aqueous humor dynamics of patients with ocular hypertension undergoing medical therapy. Arch Ophthalmol. 2012 Jun;130(6):677-84. doi: 10.1001/archophthalmol.2011.2573. PMID 22332206

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient who was taking latanoprost for ocular hypertension did not have an IOP rise greater than 20mmHg after discontinuing treatment for up to 12 weeks. A second patient who initially expressed interest chose to withdraw from the study.
Groups:
- Latanoprost/Timolol/Dorzolamide; Dorzolamide/Latanoprost/Timolol; Dorzolamide/Timolol/Latanoprost; Timolol/Dorzolamide/Latanoprost; Timolol/Latanoprost/Dorzolamide: The participants received latanoprost at night and vehicle in the morning for two weeks, then 6 week washout, then Dorzolamide BID for two weeks, then 6 week washout, then Timolol BID for two weeks. The order in which the participants received the three different drugs was random.
Period: First Intervention
Arm/Group | Latanoprost/Dorzolamide/Timolol | Latanoprost/Timolol/Dorzolamide | Dorzolamide/Latanoprost/Timolol | Dorzolamide/Timolol/Latanoprost | Timolol/Dorzolamide/Latanoprost | Timolol/Latanoprost/Dorzolamide
Started | 4 | 4 | 5 | 5 | 5 | 5
Completed | 4 | 4 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Latanoprost/Dorzolamide/Timolol | Latanoprost/Timolol/Dorzolamide | Dorzolamide/Latanoprost/Timolol | Dorzolamide/Timolol/Latanoprost | Timolol/Dorzolamide/Latanoprost | Timolol/Latanoprost/Dorzolamide
Started | 4 | 3 (1 participant dropped out between the first and second intervention due to car accident) | 4 (1 participant dropped out between first intervention and second intervention due to increased IOP) | 5 | 4 (1 participant dropped out between first intervention and second intervention due to increased IOP) | 5
Completed | 4 | 3 | 4 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Latanoprost/Dorzolamide/Timolol | Latanoprost/Timolol/Dorzolamide | Dorzolamide/Latanoprost/Timolol | Dorzolamide/Timolol/Latanoprost | Timolol/Dorzolamide/Latanoprost | Timolol/Latanoprost/Dorzolamide
Started | 4 | 3 | 4 | 5 | 3 (1 participant dropped out between second intervention and third intervention due to increased IOP) | 5
Completed | 4 | 3 | 4 | 5 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Latanoprost/Dorzolamide/Timolol
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Description: Intra-ocular Pressure was measured by applanation tonometry
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Latanoprost: The participants received latanoprost 0.004% at night and vehicle in the morning for two weeks
- Timolol: The participants received timolol 0.5% BID for two weeks
- Dorzolamide: The participants received dorzolamide 2% BID for two weeks
Arm/Group | Latanoprost | Timolol | Dorzolamide
Number analyzed (Participants) | 28 | 24 | 26
mmHg
  Daytime | 17.6 (3.7) | 16.4 (2.3) | 20.2 (4.8)
  Night time | 17.0 (3.2) | 17.1 (2.5) | 17.6 (2.4)
Statistical Analysis 1: Comparison: Latanoprost vs Timolol vs Dorzolamide; Test type: Equivalence — ANOVA was performed to compare the results between the three interventions; p < .05, ANOVA — threshold for significance was <0.05

2. Primary Outcome: Aqueous Flow
Description: aqueous flow measurements was calculated using fluorophotometry measurements.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: μL/min
Arm/Group | Latanoprost | Timolol | Dorzolamide
Number analyzed (Participants) | 28 | 24 | 26
μL/min
  day time | 2.09 (0.71) | 1.57 (0.44) | 1.75 (0.54)
  night time | 1.1 (0.38) | 1.1 (0.38) | 1.1 (0.38)
Statistical Analysis 1: Comparison: Latanoprost vs Timolol vs Dorzolamide; Test type: Equivalence — ANOVA was performed to compare the results between the three interventions; p < 0.05, ANOVA — threshold for statistical significance was <0.05

3. Primary Outcome: Central Corneal Thickness
Description: central corneal thickness was measured by ultrasound pachymetry
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Latanoprost | Timolol | Dorzolamide
Number analyzed (Participants) | 28 | 24 | 26
μm
  day time | 564 (40) | 568 (43) | 564 (44)
  night time | 585 (46) | 586 (45) | 582 (43)
Statistical Analysis 1: Comparison: Latanoprost vs Timolol vs Dorzolamide; Test type: Equivalence — ANOVA was performed to compare the results between the three interventions; p = 0.93, ANOVA — threshold for statistical significance was <0.05

4. Primary Outcome: Anterior Chamber Volume
Description: Anterior chamber volume was measured by A-scan ultrasound biometry, daytime
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: μL
Arm/Group | Latanoprost | Timolol | Dorzolamide
Number analyzed (Participants) | 28 | 24 | 26
μL | 191 (45) | 191 (33) | 198 (38)
Statistical Analysis 1: Comparison: Latanoprost vs Timolol vs Dorzolamide; Test type: Equivalence — ANOVA was performed to compare the results between the three interventions; p = 0.84, ANOVA — threshold for statistical significance was <0.05

5. Primary Outcome: Blood Pressure
Description: blood pressure was measured by sphygmomanometry
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost | Timolol | Dorzolamide
Number analyzed (Participants) | 28 | 24 | 26
mmHg
  systolic day time | 136 (20) | 138 (22) | 139 (19)
  systolic night time | 143 (17) | 136 (15) | 138 (17)
  diastolic day time | 78 (12) | 81 (12) | 83 (11)
  diastolic night time | 83 (11) | 79 (11) | 82 (12)
Statistical Analysis 1: Comparison: Latanoprost vs Timolol vs Dorzolamide; Test type: Equivalence — ANOVA was performed to compare the results between the three interventions; p < 0.05, ANOVA — threshold for statistical significance was <0.05

6. Primary Outcome: Episcleral Venous Pressure
Description: Episcleral venous pressure was measured by venomenometry
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Latanoprost | Timolol | Dorzolamide
Number analyzed (Participants) | 28 | 24 | 26
mmHg | 9.4 (1.4) | 9.6 (1.3) | 9.4 (1.0)
Statistical Analysis 1: Comparison: Latanoprost vs Timolol vs Dorzolamide; Test type: Equivalence — ANOVA was performed to compare the results between the three interventions; p = 0.89, ANOVA — threshold for statistical significance was <0.05

7. Primary Outcome: Outflow Facility
Description: outflow facility was calculated using fluorophotometry and tonography
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: µL/min per mm Hg
Arm/Group | Latanoprost | Timolol | Dorzolamide
Number analyzed (Participants) | 28 | 24 | 26
µL/min per mm Hg
  day time fluorophotometry | 0.23 (0.18) | 0.23 (0.12) | 0.21 (0.11)
  daytime tonography | 0.22 (0.10) | 0.18 (0.08) | 0.20 (0.08)
  night tonography | 0.21 (0.11) | 0.17 (0.08) | 0.18 (0.08)
Statistical Analysis 1: Comparison: Latanoprost vs Timolol vs Dorzolamide; Test type: Equivalence — Kruskal-Wallis test was used to compare the differences between outflow facility for the three interventions; p < 0.05, Kruskal-Wallis — threshold for statistical significance was <0.05

8. Primary Outcome: Uvescleral Outflow
Description: uvescleral outflow was calulated using goldmann equation
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: µL/min per mm Hg
Arm/Group | Latanoprost | Timolol | Dorzolamide
Number analyzed (Participants) | 28 | 24 | 26
µL/min per mm Hg
  day time fluorophotometry | 0.43 (1.64) | -0.16 (1.13) | 0.14 (1.21)
  daytime tonography | 0.90 (1.46) | 0.70 (1.52) | 0.58 (1.62)
  night tonography | 0.26 (1.10) | 0.50 (1.38) | 0.12 (1.45)
Statistical Analysis 1: Comparison: Latanoprost vs Timolol vs Dorzolamide; Test type: Equivalence — Kruskal-Wallis test was used to compare the differences in uveoscleral outflow between the three interventions; p < 0.05, Kruskal-Wallis — threshold for statistical analysis was <0.05

ADVERSE EVENTS:
Groups:
- Latanoprost: The participants received latanoprost at night and vehicle in the morning for two weeks,
- Dorzolamide: Dorzolamide BID for two weeks,
- Timolol: Timolol BID for two weeks
Arm/Group | Latanoprost | Dorzolamide | Timolol
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No